CLINICAL TRIAL: NCT01632462
Title: A Prospective, Placebo Controlled, Double-Blind, Cross-over Study on the Effects of a Probiotic Preparation (VSL#3) on Metabolic Profile, Intestinal Permeability, Microbiota, Cytokines and Chemokines Expression and Other Inflammatory Markers in Pediatric Patients With Crohn's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Erasmo Miele, Assistant Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 06-2012
Record Dates: First submitted 2012-06-25; First posted 2012-07-03 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; VSL#3; probiotics; metabolic profile
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VSL#3 arm (Active Comparator): 15 patients with a diagnosis of Crohn's disease will be exposed to VSL#3 for 8 weeks
  Interventions: Drug: VSL#3
- placebo group (Placebo Comparator): 15 patients affected by Crohn's disease will be exposed to a placebo for 8 weeks
  Interventions: Drug: VSL#3

INTERVENTIONS:
Drug: VSL#3 — This investigation will be a randomized, double-blind, placebo-controlled, cross-over trial. The study will include 30 children with CD and will be articulated in 6 months as follows. These children will be randomised to a treatment group receiving for 2 months either 1-2 packet containing 900 billion bacteria/day of VSL#3 according to their weight, and a group receiving the placebo drug. Assignment to therapy or placebo will be determined according to a computer-generated randomization scheme.. At the completion of the 8 weeks, a "wash-out" period of 6 weeks will be done, when no preparation will be administered. Then each patient will be switched to the other group and followed likewise for further 8 weeks.

SUMMARY:
Background VSL#3 has been reported as an effective adjuvant therapy both in inducing and maintaining remission in pediatric patients affected by Ulcerative Colitis. In addition, it has been shown that VSL#3 is able to modulates barrier function, intestinal permeability, and innate host functions, which if altered, could have a profound impact on the state of colitis. However it is still unclear how VSL#3-induced changes in microbial composition affect the status of intestinal inflammation and no study have investigated the efficacy of VSL#3 in the maintenance of remission in pediatric patients with Crohn's disease (CD).

Objectives The purpose of this study will be to evaluate the effect of a probiotic formulation, VSL#3, versus placebo, on metabolic profile, intestinal permeability, microbiota, cytokines and chemokines expression in pediatric patients with CD in remission of disease. In addition, the efficacy of VSL#3 on the maintenance of remission will be assessed and the safety and the tolerability of the probiotic formula will be evaluated.

Methods This investigation will be a prospective, multicenter, randomized, double-blind, placebo-controlled, cross-over trial. The study will include 50 children affected by CD in remission of disease, as defined by a PCDAI < 10, under treatment with Azathioprine associated or not to 5-ASA and will be articulated in 6 months as follows. All children will be randomised to a treatment group receiving for 2 months either 1-2 packet containing 900 billion bacteria/day of VSL#3 according to their weight, and a group receiving the placebo drug. Assignment to therapy or placebo will be determined according to a computer-generated randomization scheme. At the completion of the 8 weeks, a "wash-out" period of 6 weeks will be done, when no preparation will be administered. Then each patient will be switched to the other group and followed likewise for further 8 weeks. All patients will continue regular medications throughout the study period. A group of 10 volunteer healthy children, comparable in age and sex, will be used as reference group for the analysis of metabolic profile. Patients will be assessed clinically at baseline and every 8 weeks until the completion of the study, at 24 weeks or at the time of relapse. At every visit data will be collected including patient questionnaires regarding disease activity (stool frequency, stool consistency, hematochezia, abdominal pain, extraintestinal manifestations of disease, and overall patient functioning). Additional information collected at the first visit included demographic data, family history, and symptom onset. Physical examination will be performed at each visit by a paediatrician and included an abdominal examination and examination for extraintestinal manifestations of CD. Routine blood tests for CD, cellobiose/mannitol small intestinal permeability study, stool cultures, stool calprotectin, will be performed at every visit and/or at the time of relapse. Urine will be collected for the analysis of metabolic profile with mono and bi-dimensional high-resolution 1H NMR spectroscopy. PCDAI and a physician's global assessment will be used to measure disease activity. At baseline and at 24 weeks the patients will undergo ileocolonoscopy to evaluate and endoscopic and histological activity of disease. Evaluation of microbiota on biopsies and stool samples will be performed at the time of ileocolonoscopies using Fluorescence In Situ Hybridization. Colon biopsies cultures will be performed in order to evaluate cytokines and chemokines patterns by multiplex assay. Additional data will be collected during the study regarding the safety and tolerability of therapy with VSL #3. Statistical analysis will be performed using SPSS version 15 (SPSS Inc, Chicago, Illinois, USA). Variables will be screened for their distribution and appropriate parametric or non parametric tests will be adopted as required. Cross-tabulations will be evaluated by using the Fisher test and χ2test. Statistical significance will be predetermined as P < 0.05.

Expected results The investigators expect to find profound alterations in metabolic profiles, intestinal permeability, microbiota, cytokines and chemokine patterns of patients affected by CD. The administration of VSL#3 is expected to ameliorate all these alterations eventually identified. From a clinical point of view the effects of VSL#3 could be translated in prolonged clinical remission maintenance, offering a new therapeutic tool in the treatment of CD.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD) in childhood are chronic relapsing and remitting inflammatory condition that have a significant impact on growth and development.

IBD involves a shift from a regulated intestinal immune response to one that is driven by unrestrained immune cell activation and pro-inflammatory cytokine production. (1) The cause of this increase in immune stimulation is of great interest and several studies indicate a role for commensal bacteria in the progression of disease. (2) A recent study compared the microbiota of patients with IBD with that of non-IBD controls and revealed a significant difference in their composition. The microbiota of IBD patients showed abnormal microbial composition characterized by depletion of Firmicutes and Bacteroides, which are represented in non-IBD controls. (3)

Enhanced NF-κB activity is involved in the pathology of both forms of IBD. Crohn disease (CD) and ulcerative colitis (UC). The mechanism of proteasome-mediated NF-κB activation in CD and UC has been studied. Visekruna et al demonstrated that the subunit composition and the proteolytic function of proteasomes differ between UC and CD. High expression of the immunoproteasome subunits β1i and β2i is characteristic of the inflamed mucosa of CD (4). In line with this, they found enhanced processing of NF-κB precursor p105 and degradation of inhibitor of NF-κB, IκBα, by immunoproteasomes isolated from the mucosa of CD patients. In comparison with healthy controls and CD patients, UC patients exhibited an intermediate phenotype regarding the proteasome-mediated processing/degradation of NF-κB components (4) .Finally, increased expression of the NF-κB family member c-Rel in the inflamed mucosa of CD patients suggests that p50/c-Rel is important for IFN-γ-mediated induction of immunoproteasomes via IL-12-driven Th1 responses. These findings suggest that distinct proteasome subunits influence the intensity of NF-κB-mediated inflammation in IBD patients (4).

In the study of Pagnini C et al., the authors report that the probiotic mixture VSL#3 prevents the onset of intestinal inflammation in the SAMP mouse model of CD-ileitis. These effects were associated with a local effect on the intestinal epithelium (i.e., stimulation of TNF-α production and NF-κB activation in epithelial cells, coupled with restitution of normal intestinal epithelial barrier function).

Analysis of bacterial DNA in the stool and ileal mucosa of treated mice demonstrated a significant increase of probiotic strains, suggesting that effective bacterial colonization is required for the beneficial effects of probiotic treatment. This study support the hypothesis that probiotics promote gut health through a mechanism involving stimulation of epithelial innate responses (i.e., stimulation of TNF-α expression), rather than suppression of inflammation. (5)

Many individual or combinations of bacterial species have been shows to ameliorate the symptoms of IBD and to reduce intestinal inflammation in animal studies. Treatment of mice with colitis with the probiotic formulation VSL#3 increased the production of IL-10 and the percentage of TGFβ-expressing T-cells. Transfer of lamina propria mononuclear cells from VSL#3-treated mice prevented colitis in recipient mice, indicating that the VSL#3 can initiate the generation of a protective population of cells. (6)

The recent identification of symbiotic bacteria with potent anti-inflammatory properties, and their correlative absence during disease, suggests that certain aspects of human health may depend on the status of microbiota. (7)

In addition, the Lipopolysaccharide (LPS) is a major component of the bacterial outer membrane that is largely responsible for mediating septic shock. Normally the body does not react to the high concentration of LPS that is present in the intestinal lumen. Intestinal alkaline phosphatase (IAP) seems to detoxify LPS by hydrolyzing it and maintaining intestinal homeostasis with the commensal flora. (8)

Probiotics modulate the composition of the gut microbiota. Global microarray and bioinformatica analysis revealed augmentation of immune response, phagocytic, and inflammatory pathways dominated by elevation of Th1 transcription factors in IL10-KO mice. IL10-KO mice orally administered with the probiotic VSL#3 exhibited a site-specific downregulation of these inflammatory pathways including TLR signalling and related effector pathways such as T-cell, B-cell receptor signaling. More important, VSL#3 triggered an up-regulation in PPAR signaling, lipid, nitrogen, amino acid, and xenobiotic metabolism (9).

Actually it is unclear how VSL#3-induced changes in microbial composition affect the status of intestinal inflammation. It is possible that VSL#3 promotes the presence of protective microorganisms, likely constituents of the probiotic itself that directly influence host innate responses. It has been reported that VSL#3 modulates barrier function, intestinal permeability, and innate host functions, which if altered, could have a profound impact on the state of colitis. VSL#3 has been shown to enhance barrier function through decreased epithelial permeability in IL10_/_ mice, correlating with a reduction in intestinal inflammation. Another recent study demonstrated that VSL#3 prevents the development of ileitis in SAMP1/YitFc mice by enhancing epithelial barrier function and activating innate signaling leading to NF-jB activation. These effects appear to be mediated by VSL#3 secreted products. This is consistent with reports showing that probiotic-derived factors are capable of modulating host responses and experimental colitis. Additionally, structural components present in probiotic bacteria could profoundly impact immune response and favor the production of immunosuppressive molecules such as IL-10 (10).

Purpose:

The purpose of this study is to evaluate the effect of a probiotic formulation, VSL#3, versus placebo, on metabolic profile, intestinal permeability, microbiota, cytokines and chemokines expression and other inflammatory markers in pediatric patients with Crohn's Disease (CD) in remission (11).

Secondary objectives are:

* To determine the effect on Pediatric Crohn Disease Activity Index (PCDAI)
* to determine the time till flare of CD pediatric patients on VSL#3 compared to placebo
* to assess whether concurrent therapy with VSL#3 reduces the severity of a flare if it occurs
* to assess the safety and tolerability of therapy with VSL #3 at high dosage in pediatric patients with CD

Study design

This investigation will be a randomized, double-blind, placebo-controlled, cross-over trial. The study will include 30 children with CD and will be articulated in 6 months as follows. A group of 10 volunteer healthy children, comparable in age and sex, will be used as reference group for the analysis of metabolic profile..

These children will be randomised to a treatment group receiving for 2 months either 1-2 packet containing 900 billion bacteria/day of VSL#3 according to their weight, and a group receiving the placebo drug. Assignment to therapy or placebo will be determined according to a computer-generated randomization scheme. The medications will be dispensed by the investigator at each visit; compliance will be assessed by counting returned bags and questioning the patients. Excellent compliance will be defined as no violation of the protocol with respect to the intake of the study medication. At the completion of the 8 weeks, a "wash-out" period of 6 weeks will be done, when no preparation will be administered. Then each patient will be switched to the other group and followed likewise for further 8 weeks.

All patients will continue regular medications throughout the study period (azathioprine associated or not to 5-ASA).

Patients will be assessed clinically at baseline and every 8 weeks until the completion of the study, at 24 weeks or at the time of relapse. At every visit data will be collected including patient questionnaires regarding disease activity (stool frequency, stool consistency, hematochezia, abdominal pain, extraintestinal manifestations of disease, and overall patient functioning). Additional information collected at the first visit included demographic data, family history, and symptom onset. Physical examination will be performed at each visit by a paediatrician and included an abdominal examination and examination for extraintestinal manifestations of CD. Routine blood tests for CD, cellobiose/mannitol small intestinal permeability study, stool cultures, stool calprotectin, will be performed at every visit and/or at the time of relapse. Urine will be collected for the analysis of metabolic profile with mono and bi-dimensional high resolution 1H NMR spectroscopy. In 10 healthy volunteer children and patients, bile acid, isoleucine, leucine, valine, 2-oxo-3methyl-valeric acid, 2-oxo-isovaleric acid, 2-methyl-3-hydroxybutyric acid, 3-hydroxybutyrate, 3-hydroxybutyrate, 3-hydroxyisovaleric acid, threonine, lactate, 3-hydroximethylglutamic acid, alanine, N-acetyl asparagine + aspartyl glutamate + glutamil acid, acetic acid, carnitine, acetone, acetoacetate, 2-hydroxyglutarate, pyruvate, glutaric acid, N-Acetylglutamic acid, succinate, 3-hydroxy-3-methylglucaric acid, dimethylamine, sarcosine, N-acetyl-aspartyl-glutamate, dimethylglycine, citric acid, creatine, creatinine, choline, betaine, malonic acid, trimethylamineoxide, sarcosine, glycine, 1-methylhistidine, 3-methylhistidine, benzoilglycine (hippuric acid) , N-methyl betaine (trigonellina), arabinosio, uracil, guanosine, tyrosine, phenylalanine, xanthine, hypoxanthine, 3-methylhistidine will be evaluated. In addition, in children with CD, many other metabolites signals will be expected, resulting from drugs or other compounds taken as such or processed by the body's metabolism or intestinal microbial flora. the metabolomic analysis will allow the evaluation of the following organ specific and systemic processes based on low molecular weight compounds providing a profile of the metabolic system of the subjects: intermediary metabolism of sugar, mitochondrial citric acid cycle, amino acids metabolism, oxidative metabolism of fatty acid, break down and turnover of proteins, metabolism of purine and pyrimidine, pathway of trans-methylation and trans-sulphide, metabolism of intestinal bacteria; etc.

PCDAI and a physician's global assessment were used to measure disease activity. No disease activity equals a score of 0-10, mild disease equals 11-30, moderate/severe disease equals 31 or more. (10)

At baseline and at 24 weeks the patients will undergo ileocolonoscopy to evaluate and endoscopic and histological activity of disease. Evaluation of microbiota on biopsies and stool samples will be performed at the time of ileocolonoscopies using FISH (Fluorescence In Situ Hybridization). A colon culture will be performed in order to evaluate all cytokines and chemokines by multiplex assay. In addition, the RNA analysis from biopsies will be performed for the study of proteasome subunits or other inflammatory markers

Additional data will be collected during the study regarding the safety and tolerability of therapy with VSL #3.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CD as defined by clinical, radiological, histological and endoscopic criteria with negative stool culture
* Males and Females ages 5-17 years
* Subjects should have CD in remission as defined by a PCDAI < 10
* Absence of extraintestinal manifestations
* Patients receiving the following treatment:
* Azathioprine: if the dose remained constant for 8 weeks prior to the screening visit and had been used continuously for 12 weeks before screening associated or not to 5ASA: if the dose remained constant for 4 weeks before the screening visit and had been used continuously for 8 weeks before screening
* Written informed consent by parents

Exclusion Criteria:

* Patients with Ulcerative Colitis (UC)
* Subjects with documented intestinal stricture, stenosis, obstruction, fistula, abscess, ileostomy
* Patients with perianal or active CD
* Treatment with anti-TNFα, ciprofloxacin, metronidazole, systemic corticosteroids, infliximab within 12 weeks of the start of the trial
* Patients with systemic or intestinal infection
* Renal, hepatic, haematological, pulmonary, cardiac, neurologic or cerebral diseases
* Probiotic use in the previous 2 months
* Inability or unwillingness to give an informed consent
* Subjects who require outpatient antibiotic therapy.
* Patients who require surgery for complications related to CD.
* Concurrent participation in an investigational drug trial
* Documented history of allergic reaction to Lactobacillus or other probiotic compound
* Use of Lactobacillus, Bifidobacterium, Enterococcus, Saccharomyces, or any other probiotic bacterial supplement within the past 10 days
* History of endocarditis, rheumatic valvular disease, congenital cardiac malformations, or cardiac surgery
* Presence of any other significant medical condition
* Pregnant or breastfeeding female subjects

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
to evaluate the effect of a probiotic formulation, VSL#3, versus placebo, on metabolic profile, intestinal permeability, microbiota, cytokines and chemokines expression and other inflammatory markers in pediatric patients with Crohn's Disease | 22 weeks from the enrollment
  Evaluation of metabolic profile, intestinal permeability, microbiota, cytokines and chemokines expression and other inflammatory markers in pediatric patients with Crohn's before and after the exposure to VSL3 to underline any differences

SECONDARY OUTCOMES:
To determine the effect on Pediatric Crohn Disease Activity Index (PCDAI); | 8, 14, 22 weeks from the enrollment
to determine the time till flare of CD pediatric patients on VSL#3 compared to placebo. | 8, 14, 22 weeks from the enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Erasmo Miele, Assistant Professor, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy, Italy

REFERENCES:
- [Background] Elson CO, Cong Y, Weaver CT, Schoeb TR, McClanahan TK, Fick RB, Kastelein RA. Monoclonal anti-interleukin 23 reverses active colitis in a T cell-mediated model in mice. Gastroenterology. 2007 Jun;132(7):2359-70. doi: 10.1053/j.gastro.2007.03.104. Epub 2007 Apr 13. PMID 17570211
- [Background] Sartor RB. The influence of normal microbial flora on the development of chronic mucosal inflammation. Res Immunol. 1997 Oct-Dec;148(8-9):567-76. doi: 10.1016/s0923-2494(98)80151-x. No abstract available. PMID 9588836
- [Background] Frank DN, St Amand AL, Feldman RA, Boedeker EC, Harpaz N, Pace NR. Molecular-phylogenetic characterization of microbial community imbalances in human inflammatory bowel diseases. Proc Natl Acad Sci U S A. 2007 Aug 21;104(34):13780-5. doi: 10.1073/pnas.0706625104. Epub 2007 Aug 15. PMID 17699621
- [Background] Visekruna A, Joeris T, Schmidt N, Lawrenz M, Ritz JP, Buhr HJ, Steinhoff U. Comparative expression analysis and characterization of 20S proteasomes in human intestinal tissues: The proteasome pattern as diagnostic tool for IBD patients. Inflamm Bowel Dis. 2009 Apr;15(4):526-33. doi: 10.1002/ibd.20805. PMID 19067411
- [Background] Pagnini C, Saeed R, Bamias G, Arseneau KO, Pizarro TT, Cominelli F. Probiotics promote gut health through stimulation of epithelial innate immunity. Proc Natl Acad Sci U S A. 2010 Jan 5;107(1):454-9. doi: 10.1073/pnas.0910307107. Epub 2009 Dec 14. PMID 20018654
- [Background] Di Giacinto C, Marinaro M, Sanchez M, Strober W, Boirivant M. Probiotics ameliorate recurrent Th1-mediated murine colitis by inducing IL-10 and IL-10-dependent TGF-beta-bearing regulatory cells. J Immunol. 2005 Mar 15;174(6):3237-46. doi: 10.4049/jimmunol.174.6.3237. PMID 15749854
- [Background] Round JL, Mazmanian SK. The gut microbiota shapes intestinal immune responses during health and disease. Nat Rev Immunol. 2009 May;9(5):313-23. doi: 10.1038/nri2515. PMID 19343057
- [Background] Geddes K, Philpott DJ. A new role for intestinal alkaline phosphatase in gut barrier maintenance. Gastroenterology. 2008 Jul;135(1):8-12. doi: 10.1053/j.gastro.2008.06.006. Epub 2008 Jun 10. No abstract available. PMID 18549817
- [Background] Reiff C, Delday M, Rucklidge G, Reid M, Duncan G, Wohlgemuth S, Hormannsperger G, Loh G, Blaut M, Collie-Duguid E, Haller D, Kelly D. Balancing inflammatory, lipid, and xenobiotic signaling pathways by VSL#3, a biotherapeutic agent, in the treatment of inflammatory bowel disease. Inflamm Bowel Dis. 2009 Nov;15(11):1721-36. doi: 10.1002/ibd.20999. PMID 19639558
- [Background] Uronis JM, Arthur JC, Keku T, Fodor A, Carroll IM, Cruz ML, Appleyard CB, Jobin C. Gut microbial diversity is reduced by the probiotic VSL#3 and correlates with decreased TNBS-induced colitis. Inflamm Bowel Dis. 2011 Jan;17(1):289-97. doi: 10.1002/ibd.21366. PMID 20564535
- [Background] Hyams JS, Ferry GD, Mandel FS, Gryboski JD, Kibort PM, Kirschner BS, Griffiths AM, Katz AJ, Grand RJ, Boyle JT, et al. Development and validation of a pediatric Crohn's disease activity index. J Pediatr Gastroenterol Nutr. 1991 May;12(4):439-47. PMID 1678008